CLINICAL TRIAL: NCT00339287
Title: Molecular Basis of Human Phagocyte Interactions With Bacterial Pathogens
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901055; 01-I-N055
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-07-08

CONDITIONS: Host Defense Mechanisms
Keywords: Virulence; PHAGOCYTOSIS; Neutrophil; Pathogenesis; Natural History

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers: Healthy adult volunteers at least 18 years of age.

SUMMARY:
Human phagocytic cells such as polymorphonuclear leukocytes (PMNs) are readily mobilized to sites of infection and ingest microorganisms by a process known as phagocytosis. The combined effects of reactive oxygen species (ROS) and proteolytic peptides and enzymes released into forming bacterial phagosomes kill most ingested bacteria. However, many human bacterial pathogens have devised means to subvert normal phagocyte responses and the innate immune response and cause severe disease.

The overall objective of this study is to elucidate specific features of pathogen-phagocyte interactions that underlie evasion of the innate immune response or contribute to the pathophysiology of disease or inflammatory disorders. Therefore, specific projects will:

1. Identify and characterize specific mechanisms used by pathogenic microorganisms to evade or subvert normal phagocyte responses and therefore cause disease.
2. Investigate phagocyte response mechanisms to specific pathogenic microorganisms.
3. Identify specific bacterial structures and/or (gene) products that dictate differences in phagocyte responses among a range of pathogens so that generalized statements can be made about the pathophysiology of disease states.

The studies will be performed using multiple techniques including state-of-the-art equipment for genomics and proteomics strategies to identify target bacterial genes/proteins of interest or those up-regulated in phagocytes. Phagocyte-pathogen interactions will be examined using fluorescence-based real-time assays and video microscopy, confocal and electron microscopy in combination with enzymatic assays for ROS production, routine biochemistry, immunology and cell biology.

Implementing these studies will require isolation of phagocytic leukocytes from venous blood of healthy human volunteers. The study population will be all-inclusive except in certain instances where individuals possess genetic defects that impair phagocyte function (e.g., myeloperoxidase-deficiency) or have altered phagocyte function due to outside influences such as recent bacterial or viral infection.

The proposed studies will likely provide new information pertinent to understanding host cell-pathogen interactions and the pathophysiology of inflammatory conditions.

DETAILED DESCRIPTION:
Human phagocytic cells such as polymorphonuclear leukocytes (neutrophils or PMNs) are readily mobilized to sites of infection and ingest microorganisms by a process known as phagocytosis. The combined effects of reactive oxygen species (ROS) and antimicrobial peptides released into forming bacterial phagosomes kill most ingested bacteria. However, many bacterial pathogens have devised means to evade normal phagocyte responses and cause severe disease in humans.

The overall objective of this study is to elucidate specific features of pathogen-phagocyte interactions that underlie evasion of the innate immune response or contribute to the pathophysiology of disease or inflammatory disorders. Therefore, projects will address 3 specific aims:

1. Identify and characterize specific mechanisms used by pathogenic microorganisms to evade or subvert normal phagocyte responses and therefore cause disease.
2. Investigate phagocyte response mechanisms to specific pathogenic microorganisms.
3. Identify specific bacterial structures and/or (gene) products that dictate differences in phagocyte responses among a range of pathogens so that generalized statements can be made about the pathophysiology of disease states.

The studies will be performed using multiple techniques including state-of-the-art equipment for genomics and proteomics strategies to identify target bacterial genes/proteins of interest or those up-regulated in phagocytes. Phagocyte-pathogen interactions will be examined using fluorescence-based real-time assays and video microscopy, confocal and electron microscopy in combination with enzymatic assays for ROS production, routine biochemistry, immunology and cell biology.

Implementing these studies will require isolation of phagocytic leukocytes from venous blood of healthy human volunteers. The study population will be all-inclusive except in certain instances where individuals possess genetic defects that impair phagocyte function (e.g., myeloperoxidase-deficiency) or have altered phagocyte function due to outside influences such as recent bacterial or viral infection.

The proposed studies will likely provide new information pertinent to understanding host cell-pathogen interactions and the pathophysiology of inflammatory conditions.

ELIGIBILITY:
* INCLUSION & EXCLUSION CRITERIA:

Volunteers will be selected from a healthy adult population, 18 years of age or older, with no known medical problems and will generally be NIH employees working at Rocky Mountain Laboratories (RML) or within the community of Hamilton, MT.

No race or gender is excluded from the donor pool and reflects the diversity of the community and that of the employees at RML.

The specific criteria for eligibility are as follows:

* Subjects must fit the definition of "healthy adults" as assessed by the medical/health screening evaluations, and willing to have blood and/or tissue samples stored for future use.
* Inasmuch as all subjects are RML employees, they will be 18 years of age or older.
* Children are excluded.
* Pregnant women will be identified by verbal history and are not eligible to donate blood for this protocol.
* The study population will be all-inclusive except in certain instances where individuals possess genetic defects that impair phagocyte function (e.g., myeloperoxidase-deficiency) or have altered phagocyte function due to outside influences such as recent bacterial or viral infection.
* Individuals below the normal hematocrit and hemoglobin ranges will be excluded from the protocol.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers will be selected from a healthy adult population, 21-65 years of age, with no known medical problems and will generally be NIH employees working at Rocky Mountain Laboratories (RML) or within the community of Hamilton, MT. No race or gender is excluded from the donor pool and reflects the diversity of the community and that of the employees at RML.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2001-02-12 (Actual)

PRIMARY OUTCOMES:
identify and characterize specific mechanisms used by pathogenic microorganisms to evade or subvert normal phagocyte responses and therefore cause disease. | Ongoing
  The study involves the use of human subjects as a source of blood for in vitro assays with bacteria, the isolation of hematopoietic cells (polymorphonuclear leukocytes, mononuclear phagocytes, erythrocytes, and lymphocytes), and serum as a source of complement, antibody, and matrix-binding proteins.

CONTACTS AND LOCATIONS:
Overall Officials: Frank R De Leo, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- NIAID, Rocky Mountain Laboratories, Hamilton, Montana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rungelrath V, DeLeo FR. Staphylococcus aureus, Antibiotic Resistance, and the Interaction with Human Neutrophils. Antioxid Redox Signal. 2021 Feb 20;34(6):452-470. doi: 10.1089/ars.2020.8127. Epub 2020 Jun 23. PMID 32460514
- [Background] Kobayashi SD, Malachowa N, DeLeo FR. Neutrophils and Bacterial Immune Evasion. J Innate Immun. 2018;10(5-6):432-441. doi: 10.1159/000487756. Epub 2018 Apr 11. PMID 29642066